CLINICAL TRIAL: NCT02933788
Title: Effect of aSpirin Versus CilOstazol for Inhibition of Antiplatelet aggRegaTion in Type 2 DM Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kangbuk Samsung Hospital (Other)
Collaborators: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hyun Kim, Fellowship, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ESCORT_DM
Record Dates: First submitted 2016-09-18; First posted 2016-10-14 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: cardiovascular disease; atherosclerosis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Atherosclerosis | interventions — Cilostazol; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cilostazol group (Experimental): Cilostazol Cilostazol 200mg tablet by mouth, once daily for 14 days
  Interventions: Drug: Cilostazol
- Aspirin group (Active Comparator): Acetylsalicylic acid Acetylsalicylic acid 100mg tablet by mouth, once daily for 14 days
  Interventions: Drug: Acetylsalicylic acid

INTERVENTIONS:
Drug: Cilostazol — Cilostazol sustained release capsule is new drugs developed by Otsuka Korea. This drugs have platelet aggregation inhibiting action, peripheral vasodilating action and endothelial function improving action.
  Other Names: Pletal
  Arms: Cilostazol group
Drug: Acetylsalicylic acid — Aspirin may prevent coronary thrombosis in patients with cardiovascular event risk factors, such as ischemic heart disease family history, hypertension, diabetes mellitus, dyslipidemia and obesity.
  Other Names: Aspirin
  Arms: Aspirin group

SUMMARY:
This study evaluates the more suitable treatment for the prevention of vascular complications in diabetes patents who were at high cardiovascular risk group by comparing the platelet aggregation inhibitory effect of aspirin and cilostazol.

DETAILED DESCRIPTION:
Diabetes is a dangerous disease with high risk of vascular complications. Thus, to prevent these vascular complication, antithrombotic drug may be administered. Representative antithrombotic agents are aspirin and cilostazol. However, recent studies suggested that aspirin did not have sufficient effect to prevent vascular complications of diabetes. For that reason, it have been reported that antithrombotic effects of aspirin were falling in diabetes patients, so-called 'aspirin resistance.

On the other hand, cilostazol used as the control drug inhibits atherosclerosis in diabetes patients in the studies of Asia including Korea, and it is effective to inhibit the risk of various cardiovascular disease. Therefore, cilostazol is likely to use drugs as substitute for aspirin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Who have one more following risk factor:

  * Family history of cardiovascular disease
  * Hypertension
  * Smoking History
  * Dyslipidemia
  * Albuminuria
* Who do not have high risk of bleeding
* Who stop taking Cilostazol or Aspirin before randomized period 1months or
* Who have never taken the drugs

Exclusion Criteria:

* Type 1 diabetes mellitus, gestational diabetes
* Who with history of macrovascular complication including cardiovascular disease, cerebrovascular disease and peripheral vascular disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2016-10; Primary Completion 2016-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
platelet reactivity testing | Change from Baseline 'platelet reactivity testing(Aspirin reaction units and platelet function testing-100) at 14 days
  Blood sampling is collected at baseline and after taking each drugs 14 days, in the fasting state . The rate of Aspirin reaction units(ARU) change compared baseline is measured through Verify Now. The rate of platelet aggregation(seconds) dut to collagen, epinephrine was compared through the platelet function testing-100.
  1. Verify Now(ARU): It is a test developed to monitor the platelet aggregation inhibitory effects of anti-platelet drugs which used to prevent thrombosis and relapse it. By measuring the light transmission change, it outputs result to the aspirin response units(ARU)
  2. Platelet function testing-100: platelet function analyser The cartridge membrane is coated by collagen as initial matrix for platelet adhesion. When platelet adhere to the collagen, it takes place the first physical stimulation. Then, another membrane component, Adenosine diphosphate induces platelet aggregation. The analysis equipment is measuring CT(closing time) in seconds.

SECONDARY OUTCOMES:
Observation of Clinical laboratory data(total cholesterol, HDL, LDL and triglyceride | Change from baseline "total cholesterol, HDL, LDL and triglyceride, hsCRP, cluster of designation antigen 40, ligand, Dipeptidyl peptidase-4 enzyme activity, total and active glucagon like peptide-1' at 14 days.
  The rate of lipid profile(total cholesterol, HDL, LDL and triglyceride) change which is cardiovascular risk factors and diabetes mellitus complication indicators change are measured at baseline and after taking each drugs for 14 days. Thus, the effect of each drugs preventing complication in patients with diabetes mellitus may be analyzed.
  - total cholesterol(mg/dL)/ HDL(mg/dL)/ LDL(mg/dL)/ triglyceride(mg/dL)/ hsCRP(mg/dL)/ cluster of designation antigen 40(mg/dL)/ Dipeptidyl peptidase-4 enzyme activity(uM/ml)/ total and active glucagon like peptide-1(pmol/l)

CONTACTS AND LOCATIONS:
Overall Officials: Cheol Young Park, Professor, Principal Investigator — Kanbuk Samsung Diabetes Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Global status report on noncommunicable diseases 2010
- [Background] Emerging Risk Factors Collaboration; Sarwar N, Gao P, Seshasai SR, Gobin R, Kaptoge S, Di Angelantonio E, Ingelsson E, Lawlor DA, Selvin E, Stampfer M, Stehouwer CD, Lewington S, Pennells L, Thompson A, Sattar N, White IR, Ray KK, Danesh J. Diabetes mellitus, fasting blood glucose concentration, and risk of vascular disease: a collaborative meta-analysis of 102 prospective studies. Lancet. 2010 Jun 26;375(9733):2215-22. doi: 10.1016/S0140-6736(10)60484-9. PMID 20609967
- [Background] American Diabetes Association. Standards of medical care in diabetes-2015 abridged for primary care providers. Clin Diabetes. 2015 Apr;33(2):97-111. doi: 10.2337/diaclin.33.2.97. No abstract available. PMID 25897193
- [Background] Ogawa H, Nakayama M, Morimoto T, Uemura S, Kanauchi M, Doi N, Jinnouchi H, Sugiyama S, Saito Y; Japanese Primary Prevention of Atherosclerosis With Aspirin for Diabetes (JPAD) Trial Investigators. Low-dose aspirin for primary prevention of atherosclerotic events in patients with type 2 diabetes: a randomized controlled trial. JAMA. 2008 Nov 12;300(18):2134-41. doi: 10.1001/jama.2008.623. Epub 2008 Nov 9. PMID 18997198
- [Background] Kim JD, Park CY, Ahn KJ, Cho JH, Choi KM, Kang JG, Kim JH, Lee KY, Lee BW, Mok JO, Moon MK, Park JY, Park SW. Non-HDL cholesterol is an independent risk factor for aspirin resistance in obese patients with type 2 diabetes. Atherosclerosis. 2014 May;234(1):146-51. doi: 10.1016/j.atherosclerosis.2014.01.015. Epub 2014 Feb 12. PMID 24657383
- [Background] Cohen HW, Crandall JP, Hailpern SM, Billett HH. Aspirin resistance associated with HbA1c and obesity in diabetic patients. J Diabetes Complications. 2008 May-Jun;22(3):224-8. doi: 10.1016/j.jdiacomp.2007.05.002. Epub 2008 Apr 16. PMID 18413227
- [Background] Araki S, Matsuno H, Haneda M, Koya D, Kanno Y, Kume S, Isshiki K, Araki H, Ugi S, Kawai H, Kashiwagi A, Uzu T, Maegawa H. Cilostazol attenuates spontaneous microaggregation of platelets in type 2 diabetic patients with insufficient platelet response to aspirin. Diabetes Care. 2013 Jul;36(7):e92-3. doi: 10.2337/dc12-2702. No abstract available. PMID 23801816
- [Background] Henn V, Slupsky JR, Grafe M, Anagnostopoulos I, Forster R, Muller-Berghaus G, Kroczek RA. CD40 ligand on activated platelets triggers an inflammatory reaction of endothelial cells. Nature. 1998 Feb 5;391(6667):591-4. doi: 10.1038/35393. PMID 9468137
- [Background] Davi G, Catalano I, Averna M, Notarbartolo A, Strano A, Ciabattoni G, Patrono C. Thromboxane biosynthesis and platelet function in type II diabetes mellitus. N Engl J Med. 1990 Jun 21;322(25):1769-74. doi: 10.1056/NEJM199006213222503. PMID 2345567
- [Derived] Hong S, Lee WJ, Park CY. Comparative Study of Ex Vivo Antiplatelet Activity of Aspirin and Cilostazol in Patients with Diabetes and High Risk of Cardiovascular Disease. Endocrinol Metab (Seoul). 2022 Apr;37(2):233-242. doi: 10.3803/EnM.2021.1353. Epub 2022 Apr 6. PMID 35381686